CLINICAL TRIAL: NCT02933294
Title: Uniportal Versus Triportal Thoracoscopic Lobectomy and Sublobectomy for Early Stage Lung Cancer: a Multicenter Randomized Controlled Trial
Brief Title: Uniportal Versus Triportal Thoracoscopic Lobectomy and Sublobectomy for Early Stage Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other); Chinese PLA General Hospital (Other); Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Ju-Wei Mu, MD，PHD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLYXXTCX-201509
Record Dates: First submitted 2016-09-23; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Lung Neoplasms
Keywords: uniportal; lung cancer; VATS
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triportal pulmonary resection surgery (Active Comparator): Treated by traditional video assisted thoracoscopic three-port pulmonary resection in the centers with enough experience in VATS and the volume ≧50 cases each year.
  Interventions: Procedure: Triportal pulmonary resection surgery
- Uniportal pulmonary resection surgery (Active Comparator): Treated by minimally invasive video assisted thoracoscopic single-port pulmonary resection in the centers with enough experience in VATS and the volume ≧50 cases each year.
  Interventions: Procedure: Uniportal pulmonary resection surgery

INTERVENTIONS:
Procedure: Triportal pulmonary resection surgery — Uniportal video-assisted thoracoscopic surgery
  Arms: Triportal pulmonary resection surgery
Procedure: Uniportal pulmonary resection surgery — Triportal video-assisted thoracoscopic surgery
  Arms: Uniportal pulmonary resection surgery

SUMMARY:
Lung cancer is one of the most common cancers in the world. At present, surgical resection is still the standard treatment for early stage lung cancer. Triportal thoracoscopic lung resection is a routine surgically procedure for early stage lung cancer while uniportal thoracoscopic lung resection is developing rapidly in recent years. Although uniportal VATS pulmonary resection has been proven to be effective in preventing postoperative morbidities, there is still no ample evidences to demonstrate that uniportal VATS pulmonary resection is equal or superior to traditional triportal thoracoscopic pulmonary resection. The purpose of this multicenter randomized controlled trial study is to compare the uniportal VATS with traditional triportal VATS pulmonary resection in postoperative complications, long-term survival, lymph node dissection and local recurrence.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancers in the world，especially in China, where the mortality ranked first in malignant tumors whether for males or females. At present, VATS (Video-assisted thoracoscopic surgery) lobectomy is still the "gold standard" for the treatment of lung cancer. Triportal thoracoscopic lung resection is a routine surgically procedure for early stage lung cancer while uniportal thoracoscopic lung resection is developing rapidly in recent years. Retrospective study in recent years showed that the postoperative complication rate is similar between uniportal thoracoscopic surgery and triportal thoracoscopic surgery. Meanwhile, the incision is more pleasing, the inflammatory response may be milder and the hospitalization time may be shorter in the uniportal thoracoscopic surgery. But until now there is no result of the randomized controlled study on the effectiveness and the prognosis between uniportal thoracoscopic surgery and triportal thoracoscopic surgery to support this conclusion. The objective of this multicenter randomized controlled trial study is to compare the postoperative complications, long-term survival, local recurrence, other perioperative variables such as conversion rate, blood loss, lymph nodes retrieved and postoperative hospital stay between the triportal VATS pulmonary resection and uniportal VATS pulmonary resection on early stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years;
* cT1- 2N0-1M0 diagnosed by chest CT, PET-CT before operation;
* No severe comorbidity, can tolerate anesthesia;
* ECOG PS scores≤2;
* The patients sign informed consents by themselves.

Exclusion Criteria:

* Inability to tolerance of tracheal intubation and general anesthesia;
* ECOG PS scores>2;
* Severe comorbidities including: Angina occurs in 3 months, uncontrolled hypertension, Congestive heart failure, a history of myocardial infarction in 6 months before admission, severe arrhythmia, severe liver, kidney or other metabolic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative respiratory complications | 30 days after surgery
  These respiratory complications involve respiratory distress or failure after the operation with continuation of mechanical ventilation, pulmonary atelectasis requiring sputum suction by bronchoscopy, pneumonia requiring specific antibiotics confirmed by thoracic X-ray or CT scan of the thorax and a positive sputum culture, and acute respiratory distress syndrome.

SECONDARY OUTCOMES:
Blood loss | Intraoperation
  blood loss during the surgery
Lymph node dissection | Intraoperation
  During the surgery, lymph node dissection were performed. The number of removed lymph-nodes were recorded according to the postoperative pathological diagnosis, and the stations of the lymph node were recorded according to the International Association for the Study of Lung Cancer (IASLC) Lymph Node Map.
Long term survival | 5 year
  five-year survival rates after surgery
Local recurrence | 3 years
  three-year local recurrence rate after surgery
Conversion rate | Intraoperation
  conversion to thoracotomy during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Juwei Mu, MD, Principal Investigator — Collaborative Innovation Center for Cancer Medicine
Locations (4):
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Beijing Chest Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Fudan University Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided